CLINICAL TRIAL: NCT02320500
Title: Prospective Randomized Controlled Trial Comparing Conservative Therapies for the Alleviation of Knee Pain in Knee Osteoarthritis
Brief Title: Comparing Conservative Therapies for the Alleviation of Knee Pain in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Gavin Wood, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANAE-217-12; NOL 158909 (Other: Health Canada)
Record Dates: First submitted 2014-12-02; First posted 2014-12-19 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard physiotherapy (Active Comparator): Standard of care physiotherapy for knee osteoarthritis (OA) patients who have been diagnosed with knee OA and may be candidates for total knee replacement (TKA)
  Interventions: Behavioral: Standard Physiotherapy
- Myofascial-specific therapy (Experimental): Patient undergo myofascial pain-specific therapy which includes trigger point injections at the same time points as the comparator (1 session every 2 weeks for 8 weeks)
  Interventions: Other: Myofascial-specific therapy

INTERVENTIONS:
Behavioral: Standard Physiotherapy — standard of care physiotherapy once every 2 weeks for 8 weeks
  Arms: standard physiotherapy
Other: Myofascial-specific therapy — Once every 2 weeks for 8 weeks (includes trigger point injections if deemed 'necessary' by chronic pain physician)
  Arms: Myofascial-specific therapy

SUMMARY:
Patients with chronic knee pain attributed to osteoarthritis and referred to orthopedics as potential candidates for a knee replacement will receive standard physiotherapy or myofascial-specific therapy over 8 weeks. Based on the investigators pilot investigation, the investigators expect those who receive myofascial-specific therapy to experience reduced pain (compared to the standard therapy group) and increased flexibility compared to baseline levels. This simple conservative therapy could postpone (or in some cases, eliminate) the need for a knee replacement since pain is the major indication for surgery. If successful, this treatment could improve the quality of life and increase productivity for thousands suffering from knee osteoarthritis and preserve valuable health care resources.

DETAILED DESCRIPTION:
Approvals (Ethics Board and Health Canada) have already been obtained for the currently proposed prospective randomized, single-blinded, controlled clinical trial. The overall objective of the current investigation is to determine whether myofascial pain-specific therapy (which includes trigger-point injections and myofascial-specific physiotherapy) provides better pain relief and improves knee function compared to the standard-of-care physiotherapy in patients who are referred to orthopedics as potential surgical candidates. Specifically, the investigators hypotheses are that: Patients with knee osteoarthritis (OA) and who may be candidates for total knee arthroplasty 1) will have significantly reduced pain (compared to those who receive standard of care physiotherapy) and improved function (compared to baseline) with myofascial pain therapy and 2) those receiving myofascial therapy will have a delayed and/or reduced need for TKA compared to the standard-of-care physiotherapy group.

Patients with chronic knee pain attributed to osteoarthritis and referred to orthopedics as potential candidates for a knee replacement will receive standard physiotherapy or myofascial-specific therapy over 8 weeks.

The Primary outcome will be pain scores (10 point visual analogue scale (VAS)) in participants following standard-of-care physiotherapy versus myofascial pain-specific therapy for 8 weeks.

The Secondary outcomes will include:

(Comparisons between and/or within groups where appropriate):

* Pain score biweekly up to 8 weeks, at 3 months and 6 months
* Decision to proceed with surgery (yes/no)-to assess the alteration in the need for TKA
* Decision to continue treatment-(yes/no) is treatment beneficial?
* Function -Biodex, 6 min.walk test, Timed up and go- Measured at baseline and 3 months following last therapy session for standard vs. myofascial -is myofascial therapy better for function?
* Brief Pain Interference (BPI) short form- Baseline, 2 weeks and 8 weeks- to assess pain interference
* Oxford knee scores-Baseline, 2 and 8 weeks- reported functional disability (compare groups and to objective measures)
* McGill SF pain questionnaire at Baseline, 2 weeks and 8 weeks-to assess pain quality
* SF-12 at Baseline, 2 weeks and 8 weeks-to assess quality of life
* Analgesics consumed at Baseline, 2 weeks, 8 weeks, 6 months-to assess pain levels
* Compare the X-ray osteoarthritis (OA) grade with initial assessment of MTPs-Does presence of myofascial trigger points (MTPs) explain discordance between OA grade and pain?
* Pain scores on a 10 cm visual analogue scale at Baseline, 2 weeks, 6 months- assess change in pain intensity
* Surgery by 6 month follow-up? Yes/No, If so, when? - postponed or eliminated need for TKA?

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bi or unilateral knee OA
* knee pain attributed to knee OA
* referral to orthopedics as a potential candidate for knee total knee arthroplasty
* ability to comprehend/sign consent, independent mobility without assistive devices

Exclusion Criteria:

* allergy/contraindication to study medications (i.e., trigger point injections), previous knee replacement surgery
* infections of clinical abnormalities other than knee OA that could cause the knee pain
* other diagnosed chronic pain syndrome for which they are taking regular pain medications
* pregnancy or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain scores on visual analogue scale (VAS) | 8 weeks

SECONDARY OUTCOMES:
Brief pain inventory (BPI) | biweekly for 8 weeks, 3 months, 6 months
Oxford knee score | biweekly for 8 weeks, 3 months, 6 months
McGill short pain questionnaire | biweekly for 8 weeks, 3 months, 6 months
timed up and go (TUG) | Baseline, 3 months
6 minute walk test | Baseline, 3 months
Biodex functional tests | Baseline, 3 months
total knee arthroplasty? If so, when | 6 month
VAS pain scores | biweekly up to 8 weeks, then 3 months & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Henry, MD, FRCPC, Principal Investigator — Queens University/Kingston General Hospital; Gavin Wood, MD, FRCSC, Principal Investigator — Queens University/Kingston General Hospital
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada